CLINICAL TRIAL: NCT00698152
Title: A Prospective, Non-controlled, Clinical Investigation of ArComXL® Polyethylene in Total Hip Replacement
Brief Title: A Clinical Investigation of ArComXL® Polyethylene in Total Hip Replacement
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ORTHO.CR.H012
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis; Avascular Necrosis; Rheumatoid Arthritis
Keywords: Total Hip Arthroplasty; Total Hip Replacement; Hip Arthritis; Polyethylene
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ArComXL® polyethylene: ArComXL® polyethylene

SUMMARY:
The purpose of this data collection is to determine long term survival rate of ArComXL® highly cross-linked polyethylene

DETAILED DESCRIPTION:
Approximately 500 patients (cases) will be enrolled in this data collection effort and 10-year follow-up will be attempted. Follow-up will be obtained by sending a questionnaire directly to the patients by mail. The follow-up will be annually and only survivorship data will be collected.

This data collection project was developed in order to determine the actual long-term (10-year) survival rate of Biomet's ArCom XL highly cross-linked polyethylene. Data will be collated for uncemented cases only. This will eliminate the possibility of cement or cement debris being a confounding variable.

The data gathered will be collated and used to provide feedback to designing engineers, support marketing efforts, and answer potential questions from reimbursement agencies.

ELIGIBILITY:
Inclusion Criteria:

* Non inflammatory degenerative joint disease including osteoarthritis and avascular necrosis
* Rheumatoid Arthritis
* Correction of Functional Deformity
* Treatment of non-union, femoral neck fractures, trochanteric fractures of the proximal femur with head involvement, unmanageable by other techniques
* Revision of previously failed total hip arthroplasty
* Uncemented applications

Exclusion Criteria:

Absolute contraindications

* Infection, sepsis and osteomyelitis

Relative contraindications

* Uncooperative patient or patient with neurologic disorders who are incapable of following directions
* Osteoporosis
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infections which may be spread to the implant site
* Rapid joint destruction, marked bone loss, or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy or neuromuscular disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that have already made the decision to undergo Total Hip Replacement and will recieve ArComXL® polyethylene
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2006-01-23 (Actual); Primary Completion 2016-01-15 (Actual); Study Completion 2016-01-15 (Actual)

PRIMARY OUTCOMES:
Incidence of revisions and removals | Annually through 10 years
  Patient questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kacy Arnold, MBA, Study Director — Zimmer Biomet
Locations (5):
- United States (5):
  - The Orthopaedic Center, Rockville, Maryland
  - The Orthopaedic Institute of Ohio, Lima, Ohio
  - Ohio Valley Orthopedic and Sports Medicine, West Chester, Ohio
  - Scranton Orthopaedic Specialists, PC, Dickson City, Pennsylvania
  - Texas Orthopedic Specialists, PA, Grapevine, Texas